CLINICAL TRIAL: NCT05372380
Title: An Open Label, One-sequence, 3-period Study to Evaluate Drug-drug Interactions and Safety Between "BR1017-1" and "BR1017-2" in Healthy Volunteers
Brief Title: A Study to Evaluate Drug-drug Interactions Between BR1017-1 and BR1017-2 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BR-FMS-CT-119
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Hypercholesterinemia
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Atorvastatin; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequence F/AE/F+AE (Experimental): A total of 32 subjects will be enrolled in one sequence group. The investigational products (IPs) will be administered according to the treatment groups(F, AE, F+AE) assigned to on sequence group in Period 1, Period 2, and Period 3.
  Interventions: Drug: BR1017-1; Drug: BR1017-2

INTERVENTIONS:
Drug: BR1017-1 — Administration to the F/F+AE group: BR1017-1 will be administered 1 tablet QD, five-day repeat dose
  Other Names: Fimasartan 60mg
Drug: BR1017-2 — Administration to the AE group: BR1017-2 will be administered 1 tablet QD, 9-day repeat dose Administration to the F+AE group: BR1017-2 will be administered 1 tablet once QD, 5-day repeat dose.
  Other Names: Atorvastatin 40mg / Ezetimibe 10mg

SUMMARY:
To evaluate the influence of BR1017-1 and BR1017-2 on pharmacokinetics and safety when administered separately or co-administered to healthy volunteers.

DETAILED DESCRIPTION:
A total of 32 subjects will be enrolled in one sequence group. The investigational products will be administered according to the treatment groups (F, AE, F+AE) assigned to one sequence group in Period 1, Period 2, and Period 3.

ELIGIBILITY:
Inclusion Criteria:

1. Health adults aged 19 to 55 at screening.
2. Male adults whose weight is ≥50kg and female adults whose weight is ≥45kg, and their body mass index (BMI) shall be between 18.0 kg/m2 and 30.0 kg/m2 BMI (kg/m2) = weight (kg) / [height (m)]2
3. Those who are given detailed explanations about the trial and express their voluntary consent to participate in the trial by signing a written consent before screening procedure begins.

Exclusion Criteria:

1. Those who have history of clinically significant diseases including hypersensitivity reaction, intolerability and anaphylaxis to major ingredients and other ingredients of the investigational products.
2. Those who have history of clinically significant diseases related to liver (including severe hepatopathy), kidney (including severe renal impairment), digestive system (including pancreatitis), respiratory system, musculoskeletal system, endocrine system (patients with diabetic ketoacidosis, diabetic coma and precoma, type 1 diabetes, etc.), neuropsychiatric system, hemato-oncology system, cardiovascular system (including heart failure and orthostatic hypotension), etc.
3. Those who have medical history of gastrointestinal system diseases (for example: Crohn's disease, peptic ulcer disease, etc.) or operations that may influence the absorption of investigational products. (However, appendectomy, hernia operation, endoscopic polypectomy and hemorrhoids/anal fissure/anal fistula surgeries are excluded.)
4. Those who are judged unfit for the trial at screening as follows:

   * Serum ALT, AST and total bilirubin > twice the upper limit of normal levels
   * e-GFR < 60 mL/min/1.73m2 (using the CKD-EPI equation)
   * Positive to HBsAg, HCV Ab, HIV and Syphilis regain test (RPR)
   * Systolic blood pressure of > 160 mmHg or < 110 mmHg, or diastolic blood pressure of > 100 mmHg or < 70 mmHg from vital signs measured from sitting position after 3 minutes of resting.
5. Those whose test results at screening other than those mentioned in paragraph 4) above are abnormal and judged clinically significant
6. Those who have participated in other clinical trials and have been administered with other investigational products in 180 days prior to the first administration of the investigational product. (The day after the last administration of any previous clinical trial's investigational product shall be counted as day 1 of the end of trial.)
7. Those who took prescription drugs (including herbal medicine prescriptions) or OTC in 14 days prior to the first administration of the investigational products, or those who have not expressed their consent for drug prohibition from 14 days before the first administration of the investigational products until the end of study. (However, medicinal products may be administered if the subjects' safety and study results are considered to be unaffected according to the investigator's judgement.)
8. Those who have given whole blood donation in 8 weeks before the first administration of the investigational products, who have given plasma/platelet donation or received blood transfusion in 4 weeks before the first administration of the investigational products and who have not expressed their consent for blood-donation prohibition from the first administration of the investigational products until 30 days after the final administration.
9. Those who have history of continuous, excessive smoking or alcohol intake in 6 months before screening (Alcohol: > 21 units/week (1unit=10g=12.5mL); Smoking: > 10 cigarettes/day), those who cannot stop smoking or caffeine intake during hospitalization or those who cannot stop drinking from 48 hours before the first administration throughout the entire study period.

   ☞ Amount of alcohol (g) = Amount of intake (ml) x alcoholicity (%) x 0.8* (*10g=12.5mL)
10. Those who have history of diet (e.g., grapefruit juice) and health/functional food intake that can influence absorption, distribution, metabolism and excretion of the investigational products in 3 days from the first administration of the investigational product or who cannot stop the intake of such diet and food from 3 days before the first administration until the end of study.
11. Those who have drug abuse (especially centrally acting drugs including sleeping pills, centrally acting pain liver, opiates or psychoactive drugs), have history of drug abuse or whose urine drug test is positive.
12. Those who cannot use contraceptive measures (including sterilization operation of the subject and his/her partner, intrauterine contraceptive device and use of diaphragm or condom) that are allowed for clinical trials from the first administration of the investigational products until the last visit.
13. Those who have genetic problems including galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
14. Those who have history of hypersensitivity or allergy on Yellow No. 5 (Sunset Yellow FCF) ingredients.
15. Female participants who are pregnant or breastfeeding, or those whose pregnancy test is positive.
16. Others who are judged to be ineligible to participate in the trial by the investigator.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-06-04 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables - Maximum (peak) steady-state plasma drug concentration during a dosage interval(Cmax,ss) of Part A and B | 0~27 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Fimasartan alone vs. Fimasartan + Atorvastatin/ Ezetimibe) and Part B (Atorvastatin/Ezetimibe vs. Fimasartan + Atorvastatin/ Ezetimibe).
Pharmacokinetic variables - Area under the plasma concentration-time curve from time zero to time t(AUCt) of Part A and B | 0~27 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Fimasartan alone vs. Fimasartan + Atorvastatin/ Ezetimibe) and Part B (Atorvastatin/Ezetimibe vs. Fimasartan + Atorvastatin/ Ezetimibe).

SECONDARY OUTCOMES:
Pharmacokinetic variables - Time to reach maximum (peak) plasma concentration following drug administration at steady state (Tmax,ss) of Part A and B | 0~27 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Fimasartan alone vs. Fimasartan + Atorvastatin/ Ezetimibe) and Part B (Atorvastatin/Ezetimibe vs. Fimasartan + Atorvastatin/ Ezetimibe).
Pharmacokinetic variables - Minimum steady-state plasma drug concentration during a dosage interval (Cmin,ss) of Part A and B | 0~27 days after medication
  The analysis to investigate drug-drug interaction shall be divided into two parts: Part A (Fimasartan alone vs. Fimasartan + Atorvastatin/ Ezetimibe) and Part B (Atorvastatin/Ezetimibe vs. Fimasartan + Atorvastatin/ Ezetimibe).

CONTACTS AND LOCATIONS:
Overall Officials: An-Hye Kim, Principal Investigator — CHA University
Locations (1):
- CHA Bundang Medical Center, CHA University, Gyeonggi-do, Seongnam-si, South Korea